CLINICAL TRIAL: NCT05501483
Title: Adipose Tissue Heterogeneity and Its Link to Type 2 Diabetes: A Randomized Open Intervention Study That Compares Empagliflozin, Pioglitazone and Semaglutide
Brief Title: Adipose Tissue Heterogeneity and Its Link to Type 2 Diabetes
Acronym: DiaSpax
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Mikael Ryden, Professor, senior consultant, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Karolinska University Hospital; 2022-00792 and 2024-03434 (Other Grant/Funding Number: Swedish Research Council); 2021-002367-21 (EudraCT Number)
Record Dates: First submitted 2022-08-10; First posted 2022-08-15 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; empagliflozin; semaglutide

STUDY DESIGN:
Intervention Model Description: Participants are recruited to either of three groups where they receive (in addition to metformin) any of the three study drugs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pioglitazone (Active Comparator): Pioglitazone is known to affect fat cells and is used as an active comparator. It reduces HbA1c but increase fat mass slightly. We hypothesize that pioglitazone may have particular benefits in individuals with a specific adipose cellularity.
  Interventions: Drug: Pioglitazone 45 mg
- Empagliflozin (Experimental): Empagliflozin reduces HbA1c and increase lipolysis possibly due to increased glucagon secretion. It also reduces fat mass weight to a minor degree.
  Interventions: Drug: Empagliflozin 25 MG
- Semaglutide (Experimental): Semaglutide reduces body weight, including fat mass, to a more significant degree than empagliflozin but has no known direct effects on adipose tissue.
  Interventions: Drug: Semaglutide 7 MG

INTERVENTIONS:
Drug: Pioglitazone 45 mg — Starts with 45 mg
  Arms: Pioglitazone
Drug: Empagliflozin 25 MG — Starts with 25 mg
  Arms: Empagliflozin
Drug: Semaglutide 7 MG — Starts with 3 mg daily for the first 2 weeks
  Arms: Semaglutide

SUMMARY:
People with newly diagnosed type 2 diabetes treated with metformin that have not reached their HbA1c target (42-64 mmol/mol) will be recruited to the study. If they fulfill the inclusion and none of the exclusion criteria, they will be, after signing informed consent, randomized to a six-month intervention with either pioglitazone, empagliflozin or semaglutide. Fat biopsies are obtained from the subcutaneous abdominal area before and after a hyperinsulinemic-euglycemic clamp at baseline and after six months. Participants are regularly followed during this the intervention. The overall goal is to determine how antidiabetic-drugs affect white adipose tissue cellularity and whether adipose heterogeneity impacts on drug response. The primary outcome measure is the change in fat tissue lipolysis (glycerol release in isolated fat cells after hormone stimulation) before and after treatment.

DETAILED DESCRIPTION:
A detailed description of the protocol has been approved by the Swedish Medical Products Agency and the study is registered as EudraCT: 2021-002367-21.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* BMI 25 kg/m2 or higher
* HbA1c 42 mmol/mol or higher
* For fertile women, effective contraception

Exclusion Criteria:

* HbA1c 65 mmol/mol or higher
* Established cardiovascular disease and/or heart failure
* Severe psychiatric condition
* Active alcoholism
* Insulin treatment
* Anticoagulant therapy (vitamin K antagonists or equivalent)
* Pregnancy, lactation
* Positive GAD or IA2 antibodies
* Low C-peptide/glucose ratio (less than 2 measured as pmol/mg per dL)
* NT-proBNP above the upper normal reference value
* Kidney disease
* Liver disease or hepatic values over twice the upper reference value
* Severe concomitant disease including ongoing cancer

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in fat cell lipolysis after 6 months of treatment | Baseline and after six months intervention
  Change in isoprenaline-induced (over basal) lipolysis in isolated fat cells

SECONDARY OUTCOMES:
Changes in fat cell heterogeneity after 6 months of treatment | Baseline and after six months intervention
  Changes in the adiponectin/leptin mRNA expression ratio in adipose tissue measured by quantitative PCR

OTHER OUTCOMES:
Changes in tissue cellularity after 6 months of treatment (explorative outcome) | Baseline and after six months intervention
  Changes in adipose tissue cellularity measured by single-cell transcriptomic analyses of fat tissue biopsies

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
According to the ethical approval, we are not allowed to share participant data that can allow identification of the individual participants. We will present data at a group level and anonymized data in the publications that are planned to result from this study.